CLINICAL TRIAL: NCT07121257
Title: Descriptive Analysis of the Functioning of the Ventijet Mechanical Ventilator During the COVID-19 Health Crisis in Patients With Acute Respiratory Failure
Brief Title: Continuous Flow Ventilation With the Ventijet System in Acute Respiratory Distress Syndrome: a First-in-Human Feasibility and Non-Inferiority Trial
Acronym: Ventijet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Principal Investigator, Lucía Picazo Moreno, Principal Investigator and Intensive Care Specialist at Hospital del Mar, Hospital del Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ventijet01; 2020/9238 (Other: Ethics Committee for Drug Research (CEIm), Parc de Salut Mar)
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: ARDS; Mechanical Ventilation; Hypoxemic Respiratory Failure
Keywords: Continuous Flow Ventilation; Mechanical Ventilation; Jet Ventilation; VENTIJET; ARDS; Respiratory Mechanics
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Prospective, unicentric, non-randomized, single-group assignment study. All enrolled patients were initially managed with conventional mechanical ventilation (PB840) and subsequently transitioned to the Ventijet system in a sequential protocol that included predefined assessment phases (1 hour, 6 hours, 12 hours, 24 hours), followed by re-connection to conventional ventilation for additional monitoring. Each patient served as their own control.
Masking Description: No masking was applied. All investigators and clinicians were aware of the ventilation mode at each study phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Flow Ventilation with VENTIJET (Experimental): All patients were initially ventilated with a conventional mechanical ventilator (PB840) under lung-protective settings. After a 1-hour stabilization and baseline assessment period, patients were transitioned to continuous flow ventilation using the Ventijet system for up to 24 hours, followed by reconnection to the conventional ventilator for post-intervention follow-up.
  Interventions: Device: VENTIJET system

INTERVENTIONS:
Device: VENTIJET system — The Ventijet system is an investigational ventilation device delivering continuous high-velocity gas flow through a proximal nozzle. The system is designed to maintain alveolar recruitment with low driving pressures, acting as an expiratory brake. Patients received continuous flow ventilation using Ventijet for 1 to 24 hours after baseline assessment with conventional mechanical ventilation.
  Other Names: Continuous Flow Ventilation

SUMMARY:
This prospective, non-randomized, single-arm, proof-of-concept clinical trial evaluates the physiological performance and safety of the Ventijet System, a hybrid ventilation system based on continuous high-velocity gas flow. The system was conceived during the coronavirus disease 2019 (COVID-19) pandemic as a response to ventilator shortages, building upon a previously patented continuous-flow nozzle system developed by Dr. Lucas Picazo in the 1990s. The concept combines the physiological benefits of continuous flow ventilation (CFV) with the potential ease of design, monitoring, and scalability.

Patients with moderate acute respiratory distress syndrome (ARDS) - defined by a ratio of arterial partial pressure of oxygen to inspired oxygen fraction (PaO₂/FiO₂) between 150 and 200 mmHg - were first stabilized on a conventional mechanical ventilator (Puritan Bennett 840, PB840) using lung-protective settings. They were then transitioned to the Ventijet system following a structured protocol that included real-time monitoring and esophageal pressure measurements.

The primary endpoint was oxygenation, measured as the change in PaO₂ after one hour of ventilation with the Ventijet system compared to baseline values under conventional ventilation. The study was designed to demonstrate non-inferiority, with a predefined margin of ±20 mmHg in PaO₂.

Secondary outcomes included carbon dioxide clearance (PaCO₂), respiratory system mechanics, safety events, and feasibility in intensive care unit (ICU) conditions.

DETAILED DESCRIPTION:
This is a prospective, interventional, single-center clinical study conducted to evaluate the physiological effects and safety of a novel ventilation system-continuous flow ventilation with Ventijet-in adult patients diagnosed with moderate acute respiratory distress syndrome (ARDS). The objective was to compare gas exchange and pulmonary mechanics between conventional pressure-controlled ventilation and the Ventijet system, which delivers continuous flow through a high-velocity nozzle.

Ventijet is a prototype mechanical ventilator developed during the COVID-19 pandemic, motivated by the urgent need for scalable and physiologically effective ventilatory support. The system builds on the concept of continuous-flow extratracheal jet ventilation (VC-ET), originally described and patented by Dr. Lucas Picazo in the 1990s. It generates a high-speed continuous gas stream via a proximally placed nozzle (tobera), which creates an expiratory braking effect. This facilitates alveolar recruitment throughout the respiratory cycle while maintaining low airway pressures and small tidal volumes. Unlike classical jet systems, Ventijet integrates real-time safety monitoring and operates using time-cycled, volume-controlled settings, making it suitable for intensive care unit (ICU) use.

Inclusion and Exclusion Criteria

Patients were screened in the ICU and included if they met all of the following:

* Age ≥ 18 years
* Intubated and on invasive mechanical ventilation
* Diagnosis of moderate ARDS (PaO₂/FiO₂ ratio between 150-200 mmHg, Berlin definition)
* Richmond Agitation-Sedation Scale (RASS) score of -5 (deep sedation)
* Stable hemodynamic and ventilatory parameters

Exclusion criteria included:

* Obstructive pulmonary disease (e.g., chronic obstructive pulmonary disease [COPD], asthma)
* Known intracranial hypertension
* Pregnancy
* Morbid obesity (body mass index [BMI] ≥ 40 kg/m²)
* Contraindication to esophageal balloon catheter placement

Study Protocol and Ventilation Phases

All patients were first stabilized on a conventional ICU ventilator (Puritan Bennett™ 840) with lung-protective settings:

* Tidal volume ≤ 6 mL/kg predicted body weight (PBW)
* Positive end-expiratory pressure (PEEP) titrated to maintain an end-expiratory transpulmonary pressure (PLexp) between 0-2 cm H₂O
* Respiratory rate adjusted to maintain arterial pH > 7.30
* Fraction of inspired oxygen (FiO₂) adjusted to maintain oxygen saturation (SpO₂) > 92%

Once stability was confirmed, patients remained on these settings for 1 hour (Conventional-1h phase), after which a full dataset was collected, including:

* Arterial blood gas (ABG) analysis
* Respiratory and ventilatory parameters
* Hemodynamic variables
* Pulmonary mechanics

Patients were then transitioned to the Ventijet system using end-expiratory clamping to avoid alveolar derecruitment. Ventijet parameters were adjusted to approximate the previous conventional settings. After 1 hour on Ventijet (VJ-1h phase), the same dataset was recorded. This timepoint served as the primary comparison for non-inferiority analysis of oxygenation (PaO₂).

Patients who remained stable on Ventijet continued for up to 24 hours. Additional datasets were collected at 6, 12, and 24 hours (VJ-6h, VJ-12h, VJ-24h). Afterward, they were reconnected to the conventional ventilator (again using end-expiratory clamping), and evaluations were repeated at 1, 12, and 24 hours post-reconnection (Post-VJ-1h, Post-VJ-12h, Post-VJ-24h).

Monitoring and Data Collection Each study phase was supervised continuously by a trained investigator. A CARESCAPE™ B650 monitoring system (General Electric™) was used to capture ventilatory and hemodynamic parameters. Active humidification was maintained throughout. Deep sedation (RASS -5) was ensured during all Ventijet phases.

Variables collected at each phase included:

* Clinical and demographic data
* Age, sex, ICU admission diagnosis
* Comorbidities, corticosteroid use
* Neuromuscular blockers, vasoactive drugs
* Gas exchange
* Arterial partial pressures: oxygen (PaO₂), carbon dioxide (PaCO₂)
* pH, bicarbonate (HCO₃-), arterial oxygen saturation (SaO₂)
* Ventilatory variables
* Tidal volume (VT), respiratory rate (RR), PEEP
* FiO₂, inspiratory time, end-tidal CO₂ (EtCO₂), SpO₂
* Hemodynamics
* Mean arterial pressure (MAP), heart rate (HR)
* Pulmonary mechanics
* Esophageal pressure (Pes)
* Transpulmonary pressures (PLinsp, PLexp)
* Compliance of the respiratory system (Crs), lung (CL), and chest wall (Ccw)
* Driving pressures (airway and transpulmonary)

Outcomes

* Primary outcome: Change in PaO₂ between Conventional-1h and VJ-1h phases. The study was powered as a non-inferiority trial using a predefined margin of ±20 mmHg in PaO₂. Based on an estimated standard deviation of 30 mmHg, the required sample size was 14 patients (α=0.05, β=0.2).
* Secondary outcomes: Change in PaCO₂ across all phases.
* Other prespecified outcomes (collected and reported):
* Changes in respiratory mechanics (compliance, pressures)
* Duration of mechanical ventilation
* ICU and hospital length of stay
* Need for tracheostomy
* ICU, in-hospital, and 1-year mortality

Safety and Oversight

Adverse events were continuously monitored. Protocol mandated immediate reconnection to the conventional ventilator in case of:

* Hemodynamic instability
* Worsening gas exchange
* Equipment malfunction

The study was conducted in compliance with Good Clinical Practice (GCP) guidelines and was externally monitored by the Clinical Research Support Unit (SEIC) at Biocruces Bizkaia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Invasive mechanical ventilation via endotracheal tube.
* Diagnosis of moderate ARDS according to the Berlin Definition (PaO₂/FiO₂ between 150 and 200 mmHg with PEEP ≥ 5 cmH₂O).
* Lung-protective ventilation strategy prior to inclusion (VT ≤ 6 mL/kg PBW, PEEP titrated to transpulmonary pressure 0-2 cmH₂O).
* Deep sedation with RASS score of -5 at the time of inclusion.
* Informed consent obtained from the patient's legal representative.

Exclusion Criteria:

* Known obstructive pulmonary disease (e.g., COPD, asthma).
* Severe hemodynamic instability or uncontrolled shock.
* Pregnancy.
* Do-not-resuscitate (DNR) orders or limitations of life support.
* Anticipated need for ECMO in the next 24 hours.
* Presence of pneumothorax or bronchopleural fistula.
* Contraindications to esophageal pressure monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Oxygenation efficiency (PaO₂ variation at 1 hour) | 1 hour after connection to Ventijet system.
  Change in arterial partial pressure of oxygen (PaO₂) measured by arterial blood gas analysis after 1 hour of ventilation with the Ventijet system, compared to PaO₂ under conventional mechanical ventilation (PB840) after 1 hour of stabilization (conventional-1h phase).

SECONDARY OUTCOMES:
Change in arterial partial pressure of carbon dioxide (PaCO₂) after 1 hour of ventilation with VENTIJET compared to conventional ventilation. | 1 hour after connection to the Ventijet system.
  Arterial blood gas samples will be obtained after 1 hour of conventional lung-protective ventilation (conventional-1h phase) and after 1 hour of ventilation with the Ventijet system (VJ-1h phase). The primary secondary endpoint is the absolute difference in PaCO₂ between both time points. Values will be reported in mmHg.

OTHER OUTCOMES:
PaO₂/FiO₂ ratio (oxygenation index) | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Used to evaluate changes in oxygenation over time across all study phases.
PaCO₂ | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Monitored as a surrogate for CO₂ elimination efficiency during each ventilation phase.
Compliance of the respiratory system (Crs) | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Calculated using tidal volume and driving pressure to assess changes in lung mechanics with the Ventijet system vs. conventional ventilation.
Transpulmonary pressures (end-expiratory and inspiratory PL) | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Derived from esophageal pressure monitoring to evaluate lung stress and strain across phases.
Transpulmonary driving pressure (ΔPL) | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Assessed to monitor the mechanical load applied to lung parenchyma.
End-tidal CO₂ (EtCO₂) and SpO₂ | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Complementary parameters to ABG for non-invasive gas exchange monitoring.
Heart rate and mean arterial pressure (MAP) | At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.
  Hemodynamic safety endpoints.
Adverse events during Ventijet ventilation | Entire intervention and 24 hours post-Ventijet phase.
  At baseline (under conventional mechanical ventilation with PB840); after 1, 6, 12, and 24 hours of Ventijet ventilation; and at 1, 12, and 24 hours after reconnection to conventional ventilator.

CONTACTS AND LOCATIONS:
Overall Officials: Lucía Picazo, MD, Principal Investigator — Intensive Care Department, Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This was a single-center, non-randomized, proof-of-concept study with a small sample size. At present, there are no plans to share individual participant data (IPD) publicly. Data may be made available upon reasonable request and with appropriate ethical approvals.